CLINICAL TRIAL: NCT03219528
Title: A Longitudinal Study to Identify IBS Phenotypes Using Fecal Microbiota and Hydrogen Breath Testing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Michigan Institute for Clinical and Health Research (MICHR) (Unknown); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Allen Lee, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM129427; 1K23DK124567 (NIH)
Record Dates: First submitted 2017-07-13; First posted 2017-07-17 (Actual); Results first posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Diarrhea; Small Intestinal Bacterial Overgrowth; Gut Microbiota
MeSH Terms: conditions — Irritable Bowel Syndrome; Diarrhea | interventions — Rifaximin; FODMAP Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Rifaximin (Active Comparator): Rifaximin 550 mg three times daily for 14 days
  Interventions: Drug: Rifaximin 550 MG
- Low FODMAP Group (Active Comparator): Low FODMAP diet for 4 weeks
  Interventions: Other: Low FODMAP Diet

INTERVENTIONS:
Drug: Rifaximin 550 MG — Rifaximin 550 mg three times daily for 14 days
  Arms: Rifaximin
Other: Low FODMAP Diet — Low FODMAP dietary intervention for 4 weeks
  Arms: Low FODMAP Group

SUMMARY:
Diarrhea-predominant irritable bowel syndrome (IBS-D) is a highly prevalent but poorly understood condition with limited treatment options. Current therapies, including a nonabsorbable antibiotic rifaximin or diet low in fermentable oligosaccharides, disaccharides, monosaccharides, and polyols (FODMAP), show efficacy in 50% or less of patients. In this proposal, participants with IBS-D will be randomized to receive either rifaximin or low FODMAP dietary intervention.

DETAILED DESCRIPTION:
Diarrhea-predominant irritable bowel syndrome (IBS-D) is a highly prevalent but poorly understood condition with limited treatment options. Recent evidence has established small intestinal bacterial overgrowth (SIBO) and alterations in fecal microbiota as potential etiologies in the pathogenesis of IBS-D. Current therapies, including a nonabsorbable antibiotic rifaximin or diet low in fermentable oligosaccharides, disaccharides, monosaccharides, and polyols (FODMAP), show efficacy in 50% or less of patients [1-4]. It has been postulated that limited responses to therapies may stem from failure to identify distinct subgroups in IBS-D stratified by gut microbial profiles. In this proposal, participants with IBS-D will be randomized to receive either rifaximin or low FODMAP dietary intervention. The results of fecal microbiota-derived data as well as hydrogen breath tests will then be longitudinally followed to define SIBO. These methods will be used to test the hypotheses that: (i) distinct IBS-D phenotypes can be generated by defining fecal microbial populations as well as delineating the presence or absence of SIBO; and (ii) longitudinal analyses using microbe-derived metrics and SIBO status may relate to response to treatment with rifaximin or low FODMAP dietary intervention.

ELIGIBILITY:
Inclusion Criteria:

Adult subjects greater than or equal to 18 years of age who meet Rome IV criteria for diarrhea-predominant irritable bowel syndrome (IBS-D).

Prior colonoscopy or sigmoidoscopy within the past 2 years with random colon biopsies to exclude the presence of microscopic colitis.

IBS medications, including anti-depressants, will be allowed if the dose has been stable for at least 1 month before inclusion. Medications will be carefully tracked to follow any potential confounding issues.

Exclusion Criteria:

Underlying celiac disease, inflammatory bowel disease, or other organic disease that could explain their symptoms.

Subjects with a history of GI tract surgery, except for cholecystectomy or appendectomy, will also be excluded from the study.

Women who are pregnant or breastfeeding Antibiotics taken within 3 months prior to enrollment will not be permitted. Subjects on probiotics must discontinue their use at least 1 month prior to enrollment.

Subjects who have previously received formal dietary education for IBS, including a low FODMAP diet, or previously received antibiotics, including rifaximin, for treatment of IBS-D will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allen Lee, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
All investigators are aware of and agree to abide by the principles for sharing research resources, as described by NIH in "Principles and Guidelines for Recipients of NIH Research Grants and Contracts on Obtaining and Disseminating Biomedical Research Programs." The data generated in this study will be shared in several ways. Manuscripts will be submitted for publication in high-quality peer-reviewed journals. Findings will also be presented at relevant national meetings, including Digestive Disease Week and Association of Clinical and Translational Science.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rifaximin | Low FODMAP Group
Started | 38 | 36
Actual Treatment Begun | 36 | 29
Completed | 29 | 28
Not Completed | 9 | 8
Not completed — Lost to Follow-up | 5 | 4
Not completed — Withdrawal by Subject | 4 | 4

BASELINE CHARACTERISTICS:
Population: Baseline data was collected for all participants who were randomized to an arm, regardless of whether they received an intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rifaximin | Low FODMAP Group | Total
Number analyzed (Participants) | 38 | 36 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (17.9) | 44.1 (16.4) | 44.1 (17.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 26 | 56
  Male | 8 | 10 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 35 | 34 | 69
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 34 | 33 | 67
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38 | 36 | 74
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI is a medical screening tool that measures the ratio of height to weight to estimate the amount of body fat a person has.
  kg/m^2 | 29.7 (8.72) | 29.8 (8.18) | 29.8 (8.41)

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Daily Abdominal Pain
Description: Change in mean daily abdominal pain was measured using a visual analog scale (VAS) after intervention compared with baseline. VAS was a scale of 0 to 10, with higher numbers indicating a higher degree of pain; 0 indicated no pain and 10 indicated severe pain.
Time Frame: Baseline, Week 5
Population: Some participants who were randomized to an arm withdrew or were lost to follow up before receiving an intervention. The number of participants analyzed at each time point is based on a modified intent to treat (mITT) analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rifaximin | Low FODMAP Group
Number analyzed (Participants) | 36 | 29
score on a scale
  Baseline | 5.2 (1.8) | 5.3 (1.6)
  Week 5 | 3.9 (2.5) | 3.8 (2.0)
Statistical Analysis 1: Comparison: Rifaximin vs Low FODMAP Group; Baseline; Test type: Superiority; p = 0.78, Mixed Models Analysis
Statistical Analysis 2: Comparison: Rifaximin vs Low FODMAP Group; Week 5; Test type: Superiority; p = 0.88, Mixed Models Analysis

2. Secondary Outcome: Change in Irritable Bowel Syndrome (IBS) Symptom Severity Scale
Description: The IBS Symptom Severity Scale was comprised of 5 questions each of which was on a scale of 0 to 100, with higher scores indicating more severe symptoms. The total range of the scale was 0 to 500, with 0 meaning no IBS symptoms and 500 indicating severe IBS symptoms.
Time Frame: Baseline, Week 5
Population: Some participants who were randomized to an arm withdrew or were lost to follow up before receiving an intervention. The number of participants analyzed at each time point is based on a mITT analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rifaximin | Low FODMAP Group
Number analyzed (Participants) | 36 | 29
score on a scale
  Baseline | 281.3 (81.0) | 272.0 (65.1)
  Week 5 | 209.3 (81.8) | 194.7 (79.1)

3. Secondary Outcome: Change in Gastrointestinal System Ratings Scale (GSRS)
Description: The GSRS was a disease-specific instrument of 15 items combined into five symptom clusters depicting Reflux, Abdominal Pain, Indigestion, Diarrhea, and Constipation. The GSRS had a seven-point graded Likert scale where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms. The total range of the scale is 15 to 105 with 15 meaning low symptom burden and 105 meaning high symptom burden.
Time Frame: Baseline, Week 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rifaximin | Low FODMAP Group
Number analyzed (Participants) | 36 | 29
score on a scale
  Baseline | 52.0 (13.2) | 52.1 (13.3)
  Week 5 | 40.7 (11.0) | 40.1 (12.2)

4. Secondary Outcome: Change in Stool Form
Description: The Bristol Stool Form Scale was a diagnostic tool used to assess various digestive issues based on the type and shape of stool. The total range of the scale was 1 to 7, with 1 indicating hard stool and 7 indicating liquid stool.
Time Frame: Baseline, Week 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rifaximin | Low FODMAP Group
Number analyzed (Participants) | 36 | 29
score on a scale
  Baseline | 5.6 (0.8) | 5.6 (0.8)
  Week 5 | 5.0 (1.1) | 5.3 (0.9)

5. Secondary Outcome: Change in Psychological Function
Description: The PHQ-9 was a multipurpose instrument for screening, diagnosing, monitoring, and measuring the severity of depression. It is comprised of 9 questions, each ranging from 0 to 3 with higher values indicating more severe depression symptoms. The total range of the scale was 1 to 27, with 1 indicating no or minimal depression and 27 indicating severe depression.
Time Frame: Baseline, Week 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rifaximin | Low FODMAP Group
Number analyzed (Participants) | 36 | 29
score on a scale
  Baseline | 8.6 (6.5) | 8.3 (6.2)
  Week 5 | 6.2 (4.9) | 5.8 (4.3)

6. Secondary Outcome: Change in Irritable Bowel Syndrome Quality of Life Instrument (IBS-QOL)
Description: IBS-QOL was a condition-specific instrument for assessing health-related quality of life among persons with IBS. The IBS-QOL was comprised of 34 questions, each with a 5-point scale where the higher the value indicated the higher quality of life. The total range of the scale was 0 to 100, with 0 indicating no quality of life and 100 indicating extremely good quality of life.
Time Frame: Baseline, Week 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rifaximin | Low FODMAP Group
Number analyzed (Participants) | 36 | 29
score on a scale
  Baseline | 53.6 (19.5) | 58.9 (21.5)
  Week 5 | 62.6 (20.4) | 67.8 (18.5)

7. Secondary Outcome: 24-hour Diet Recall/Intake - Lactose
Description: Participants completed entries using the Nutrition Data System for Research (NDSR), which was a Windows-based dietary analysis program designed for the collection and analyses of 24-hour dietary recalls, food records, menus, and recipes. The NDSR was incapable of collecting data on all FODMAP-type foods, aside from lactose and gluten. The results represent data from lactose as a surrogate for all other FODMAP foods.
Time Frame: Baseline, Week 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: grams per day
Arm/Group | Rifaximin | Low FODMAP Group
Number analyzed (Participants) | 36 | 29
grams per day
  Baseline | 4.1 (5.5) | 7.3 (9.6)
  Week 5 | 5.1 (6.7) | 1.4 (2.3)

8. Other Pre Specified Outcome: Glucose Breath Tests
Description: Glucose breath tests (GBT) will be performed at baseline and repeated after intervention
Time Frame: 4 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Fecal Microbiota
Description: Changes in fecal microbial diversity after intervention will be compared with baseline.
Time Frame: 4 weeks
Reporting Status: Not Posted

10. Primary Outcome: Change in Mean Daily Bloating
Description: Change in mean daily bloating was measured using a visual analog scale (VAS) after intervention compared with baseline. VAS was a scale of 0 to 10, with higher numbers indicating a higher degree of bloating; 0 indicated no bloating and 10 indicated severe bloating.
Time Frame: Baseline, Week 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rifaximin | Low FODMAP Group
Number analyzed (Participants) | 36 | 29
score on a scale
  Baseline | 4.9 (1.9) | 5.1 (2.2)
  Week 5 | 4.0 (2.4) | 3.7 (2.1)
Statistical Analysis 1: Comparison: Rifaximin vs Low FODMAP Group; Baseline; Test type: Superiority; p = 0.77, Mixed Models Analysis
Statistical Analysis 2: Comparison: Rifaximin vs Low FODMAP Group; Week 5; Test type: Superiority; p = 0.58, Mixed Models Analysis

11. Secondary Outcome: 24-hour Diet Recall/Intake - Gluten
Description: Participants completed entries using the Nutrition Data System for Research (NDSR), which was a Windows-based dietary analysis program designed for the collection and analyses of 24-hour dietary recalls, food records, menus, and recipes. The NDSR was incapable of collecting data on all FODMAP-type foods, aside from lactose and gluten. The results represent data from gluten as a surrogate for all other FODMAP foods.
Time Frame: Baseline, Week 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: grams per day
Arm/Group | Rifaximin | Low FODMAP Group
Number analyzed (Participants) | 36 | 29
grams per day
  Baseline | 6.7 (6.0) | 5.7 (5.6)
  Week 5 | 7.2 (6.5) | 1.7 (4.2)

ADVERSE EVENTS:
Time Frame: 5 weeks
Description: Some participants who were randomized to an arm withdrew or were lost to follow up before receiving an intervention. The number of participants analyzed is based on a mITT analysis.
Arm/Group | Rifaximin | Low FODMAP Group
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/29
Other Adverse Events (participants affected / at risk) | 30/36 | 26/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rifaximin (N=36) | Low FODMAP Group (N=29)
Dizziness/Light-headedness (General disorders) | 1 | 0
Abdominal Pain and cramping (Gastrointestinal disorders) | 5 | 8
Bloating and gas (Gastrointestinal disorders) | 3 | 8
Heartburn (Gastrointestinal disorders) | 6 | 1
Nausea (Gastrointestinal disorders) | 5 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 5
Constipation (Gastrointestinal disorders) | 1 | 2
Headache (General disorders) | 2 | 0
Belching (Gastrointestinal disorders) | 1 | 0
Increased urination (Renal and urinary disorders) | 1 | 0
Easily sunburned (Skin and subcutaneous tissue disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Swelling (General disorders) | 1 | 0
Blurry Vision (Eye disorders) | 1 | 0
Mucus in Stool (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-06): https://cdn.clinicaltrials.gov/large-docs/28/NCT03219528/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-11): https://cdn.clinicaltrials.gov/large-docs/28/NCT03219528/ICF_002.pdf